CLINICAL TRIAL: NCT07134036
Title: Optimizing Limb Length Discrepancy in Navigated Total Hip Arthroplasty Through the Direct Anterior Approach on a Traction Table
Brief Title: Efficiency and Safety of Navigation Aids in Total Hip Arthroplasty With Direct Anterior Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Hung Hung, Division Director, China Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH112-REC1-149
Record Dates: First submitted 2025-07-05; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Hip; Femur Head Necrosis; Developmental Dysplasia of the Hip
Keywords: Direct Anterior Approach; Limb Length Discrepancy; Arthroplasty, Replacement, Hip; Surgery, Computer-Assisted; Surgical Navigation Systems
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis; Developmental Dysplasia of the Hip | interventions — Surgical Navigation Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional THA (Active Comparator): Participants in this group underwent total hip arthroplasty (THA) via the direct anterior approach on a traction table without the use of a computer navigation system. This arm represents the conventional surgical technique routinely performed at our institution, where intraoperative limb length assessment was based on standard fluoroscopic guidance and anatomical landmarks.
  Interventions: Procedure: Conventional total hip arthroplasty
- Navigation-assisted THA (Experimental): Participants in this group underwent total hip arthroplasty (THA) via the direct anterior approach on a traction table with the assistance of an imageless computer navigation system (Stryker OrthoMap Versatile Hip Navigation). The navigation system provided real-time intraoperative feedback on limb length change and acetabular cup positioning, aiming to improve accuracy and reduce reliance on fluoroscopy.
  Interventions: Device: Navigation system

INTERVENTIONS:
Device: Navigation system — Patients underwent total hip arthroplasty via the direct anterior approach using a computer navigation system to assist in intraoperative limb length measurement.
  Arms: Navigation-assisted THA
Procedure: Conventional total hip arthroplasty — Patients underwent total hip arthroplasty via the direct anterior approach conventionally.
  Arms: Conventional THA

SUMMARY:
This prospective clinical study aimed to evaluate the effectiveness of an imageless navigation system in total hip arthroplasty (THA) via the direct anterior approach (DAA) on a traction table for reducing functional limb length discrepancy (LLD) compared with conventional techniques. Seventy-two patients with advanced hip osteoarthritis, avascular necrosis, or developmental dysplasia of the hip undergoing THA between March 1, 2021 and September 30, 2021 were included. Functional LLD was assessed using a preoperative block test. Participants were assigned to the navigation or conventional group based on patient preference. Outcomes included operative parameters, intraoperative fluoroscopy time, limb length measurements, and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores.

DETAILED DESCRIPTION:
This single-center prospective comparative study was conducted at the Joint Reconstruction Center of China Medical University Hospital between March 1, 2021 and September 30, 2021. Eligible participants were adults diagnosed with advanced hip osteoarthritis, avascular necrosis, or developmental dysplasia of the hip requiring THA. Exclusion criteria included prior hip joint infection, severe LLD requiring additional reconstructive procedures, significant spinal pathology affecting spinopelvic balance, or radiographs inadequate for measurement.

All procedures were performed via the direct anterior approach (DAA) on a traction table by the principal surgeon. Functional LLD was assessed preoperatively using a block test, with wooden blocks (5 mm increments) placed under the heel until the patient reported equal leg lengths.

Patients in the navigation group underwent THA with an imageless navigation system (Stryker OrthoMap Versatile Hip Navigation) to record intraoperative limb length change and acetabular cup positioning; the conventional group underwent standard THA without navigation.

Primary outcome was the patients' expectation gap (PEG), defined as the difference between preoperative functional LLD and postoperative radiographic limb length change. Secondary outcomes included intraoperative fluoroscopy time, WOMAC scores at baseline, 3 weeks, and 3 months postoperatively, and the proportion of outliers (PEG > 10 mm).

The study was approved by the Research Ethics Committee of China Medical University Hospital (CMUH112-REC1-149). Written informed consent was obtained from all participants, and the study adhered to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced hip osteoarthritis (OA) warranting total hip arthroplasty (THA)
* Clinical diagnosis of avascular necrosis (AVN) of the femoral head warranting total hip arthroplasty (THA)
* Clinical diagnosis of developmental dysplasia of the hip (DDH) warranting total hip arthroplasty (THA)

Exclusion Criteria:

* Documented history of prior hip joint infection
* Severe limb length discrepancy requiring supplementary surgical interventions
* Significant spinal pathology affecting spinopelvic balance
* Radiographs in which the lesser trochanters and teardrops cannot be clearly defined

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Patients' Expectation Gap (PEG) | Baseline (preoperative) and 3 months postoperatively
  Difference between preoperative functional leg length discrepancy (measured with block test, mm) and postoperative radiographic leg length change (mm).

SECONDARY OUTCOMES:
Surgeons' Expectation Gap (SEG) | Intraoperative and 3 months postoperatively
  Difference between intraoperative navigation leg length measurement (mm) and postoperative radiographic leg length change (mm).
Outlier Rate (>10 mm PEG) | 3 months postoperatively
  Percentage of patients with Patients' Expectation Gap greater than 10 mm.
WOMAC Pain Score Change | Baseline, 3 weeks postoperatively, 3 months postoperatively
  Change in WOMAC pain subscale score (0-20, lower scores indicate less pain) from baseline.
WOMAC Stiffness Score Change | Baseline, 3 weeks postoperatively, 3 months postoperatively
  Change in WOMAC stiffness subscale score (0-8, lower scores indicate less stiffness) from baseline.
WOMAC Function Score Change | Baseline, 3 weeks postoperatively, 3 months postoperatively
  Change in WOMAC function subscale score (0-68, lower scores indicate better function) from baseline.
Fluoroscopy Execution Time | Intraoperative
  Duration of intraoperative fluoroscopy use (seconds).
Operative Time | Intraoperative
  Duration of total surgical procedure (minutes).
Blood Loss | Intraoperative
  Total intraoperative blood loss (milliliters).
Length Change | Baseline and 3 months postoperatively
  Difference in radiographic leg length pre- and postoperatively (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hung, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, 台中市, Taiwan

IPD SHARING:
Plan to Share IPD: No